CLINICAL TRIAL: NCT07344038
Title: Effectiveness of Bioceramic Calcium Silicate-based Pulpotomy Medicament on Primary Molars Restored With 3d Printed Resin Crowns (a Randomized Controlled Clinical Trial)
Brief Title: Bioceramic Putty Versus MTA in Pulpotomized Primary Teeth to be Covered With 3D Printed Resin Crowns Versus Stainless Steel Crown
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yousr Nader, pediatric dentistry specialist, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1155-10/2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Caries Active
Keywords: MTA, bioceramic putty, 3D printed resin crowns, stainless steel crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Endo-sequence bioceramic putty pulpotomy (Experimental)
  Interventions: Procedure: Endo-sequence bioceramic putty pulpotomy
- Bio MTA+ (Active Comparator)
  Interventions: Procedure: Bio MTA+ pulpotomy
- 3D-printed ceramic-filled hybrid resin crowns (Experimental)
  Interventions: Device: 3D-Printed Resin Crowns
- Stainless steel crowns (Active Comparator)
  Interventions: Device: Stainless Steel Crowns (SSCs)

INTERVENTIONS:
Procedure: Endo-sequence bioceramic putty pulpotomy — * Profound local anesthesia and rubber dam isolation will be applied.
  * Carious tissue will be completely removed using diamond burs until pulp exposure and deroofing.
  * Coronal pulp will be removed with a sharp excavator.
  * Hemostasis will be achieved with a saline-moistened cotton pellet for 5 minutes.
  * Bioceramic putty applied directly from the manufacturer's syringe, then adapted gently with a moist cotton pellet.
  Arms: Endo-sequence bioceramic putty pulpotomy
Procedure: Bio MTA+ pulpotomy — * Profound local anesthesia and rubber dam isolation will be applied.
  * Carious tissue will be completely removed using diamond burs until pulp exposure and deroofing.
  * Coronal pulp will be removed with a sharp excavator.
  * Hemostasis will be achieved with a saline-moistened cotton pellet for 5 minutes.
  * The MTA powder will be mixed with the liquid to a putty consistency and applied with an amalgam carrier.
  Arms: Bio MTA+
Device: Stainless Steel Crowns (SSCs) — * Occlusal reduction of 1.0-1.5 mm using a flame-shaped diamond bur.
  * Interproximal slicing to enable passive crown placement.
  * Crown size selection based on best fit.
  * Cementation using RMGIC.
  * Excess cement will be removed.
  Arms: Stainless steel crowns
Device: 3D-Printed Resin Crowns — * Tooth preparation: 1 mm axial reduction with a chamfer finish line using tapered diamond stone with round end (Mani TR-12) for buccal, lingual, mesial, and distal walls.
  * One and half - 2 mm occlusal reduction.
  * Digital impressions using IOS scanning, including occlusion and antagonist.
  * 3D printed resin crowns will be designed using the Exocad software (Exocad Rigeka 3.1) to have a uniform thickness on all surfaces (average 1 mm), including occlusal, buccal, lingual, and proximal surfaces. After reviewing each design, it will be exported as a high-resolution STL file (standard tessellation language) to be outsourced and 3D printed.
  * BEGO DLP printer will be utilized to print the crowns using VarseoSmile Trinique resin via digital light processing (DLP) technique.
  * After printing, the platform will be removed from the 3D printer and placed on a paper towel with the printed crowns facing upward.
  * The printed crowns will be separated from the platform and rinsed tw
  Arms: 3D-printed ceramic-filled hybrid resin crowns

SUMMARY:
children aged 5 to 7 years with deep carious second primary molars that require vital pulp therapy will be treated using either MTA or bioceramic putty, then will be fully covered using either stainless steel crowns or 3D printed resin crowns.

DETAILED DESCRIPTION:
removal of caries from second primary molars reaching the pulp, pulpotomy will be done by controlling the bleeding after that pulp chamber will be covered with either MTA or endosequence bioceramic putty.

resin modified glass ionomer will be placed, crown preparation will be done to receive full coverage either stainless steel crowns or 3D printed resin crowns

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 5 to 7 years. 2. Medically healthy children (ASA I) (Appendix I) 3. Positive or definitely positive behavior (Frankl's rating scale scores III or IV) (Appendix II) 4. Parents/legal guardians who provide written informed consent Tooth inclusion criteria(8, 14, 31)

  1. Deep carious second primary molars with:

     1. Vital pulp confirmed by absence of clinical and/or radiographic signs of necorosis or infection.
     2. Signs of reversible pulpitis. 10
  2. Require full coverage restorations
  3. Cooperative children (Frankl 3 or 4 behavior rating scale)

Exclusion Criteria:

* History of spontaneous pain. 2. Tooth mobility. 3. Excessive bleeding from radicular stumps after coronal pulp amputation. 4. Radiographic evidence of pathological root resorption, inter-radicular bone loss, periapical pathology, or canal calcifications. 5. Previous dental treatment of the involved molar. 6. Children with special healthcare needs.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
clinical success of pulpotomy at 1 week | clinical success at 1 week
  Clinical success: Absence of pain, sensitivity to percussion, swelling, or fistula.
clinical success of pulpotomy at 6 months | clinical success at 6 months
  Absence of pain, sensitivity to percussion, swelling, or fistula.
clinical success of pulpotomy at 12 months | clinical success at 12 months
  Absence of pain, sensitivity to percussion, swelling, or fistula.
radiographic success of pulpotomy at 1 week | radiographic success at 1 week
  No periodontal ligament space widening, resorption, or periapical/furcal radiolucency.
radiographic success of pulpotomy at 6 months | radiographic success at 6 months
  No periodontal ligament space widening, resorption, or periapical/furcal radiolucency.
radiographic success of pulpotomy at 12 months | radiographic success at 12 months
  No periodontal ligament space widening, resorption, or periapical/furcal radiolucency.
Crown evaluation at 6 months using Modified United States Public Health Service | at 6 months
  Resistance to dislodgment Alpha: Snap-fit retention Bravo: Partial retention Charlie: No retention Crown - high in occlusion Alpha: Ideal, with the crown being in harmony with occlusion.
  Bravo: Clinically acceptable, with the crown occluding slightly high or low in occlusion. Charlie: Clinically unacceptable, with the crown needing to be replaced. Retention of crown after cementation Alpha: Intact Bravo: Chipped/loss of material Charlie: Complete loss of crown Occlusal wear of crown Alpha: Occlusal surface intact. Bravo: Wear of occlusal surface without tooth surface exposure. Charlie: Wear of occlusal surface with tooth surface exposure. Wear of opposing crown or tooth Alpha: Clinically ideal, with no evidence of wear.
  Bravo: Clinically acceptable, with mild wear of the opposing tooth. Charlie: Clinically unacceptable, with severe wear of the opposing tooth. Marginal integrity and discoloration Alpha: Clinically ideal, with no evidence of gap along the gingival crown margin. Bravo: C
crown evaluation at 12 months using Modified United States Public Health Service | at 12 months
  Resistance to dislodgment Alpha: Snap-fit retention Bravo: Partial retention Charlie: No retention Crown - high in occlusion Alpha: Ideal, with the crown being in harmony with occlusion.
  Bravo: Clinically acceptable, with the crown occluding slightly high or low in occlusion. Charlie: Clinically unacceptable, with the crown needing to be replaced. Retention of crown after cementation Alpha: Intact Bravo: Chipped/loss of material Charlie: Complete loss of crown Occlusal wear of crown Alpha: Occlusal surface intact. Bravo: Wear of occlusal surface without tooth surface exposure. Charlie: Wear of occlusal surface with tooth surface exposure. Wear of opposing crown or tooth Alpha: Clinically ideal, with no evidence of wear.
  Bravo: Clinically acceptable, with mild wear of the opposing tooth. Charlie: Clinically unacceptable, with severe wear of the opposing tooth. Marginal integrity and discoloration Alpha: Clinically ideal, with no evidence of gap along the gingival crown margin. Bravo: C

SECONDARY OUTCOMES:
Parental satisfaction Assessed immediately after treatment using a 5-point Likert scale concerning appearance, color, size, durability, and overall satisfaction | immediately after treatment
  1 Very dissatisfied 2 Dissatisfied 3 Neutrally satisfied 4 Satisfied 5 Very satisfied
Parental satisfaction Assessed after 1 week using a 5-point Likert scale concerning appearance, color, size, durability, and overall satisfaction | parental satisfaction after 1 week
  1 Very dissatisfied 2 Dissatisfied 3 Neutrally satisfied 4 Satisfied 5 Very satisfied
parental satisfaction assessed after 6 months using a 5-point Likert scale concerning appearance, color, size, durability, and overall satisfaction | parental satisfaction after 6 months
  1 Very dissatisfied 2 Dissatisfied 3 Neutrally satisfied 4 Satisfied 5 Very satisfied
parental satisfaction assessed after 12 months using a 5-point Likert scale concerning appearance, color, size, durability, and overall satisfaction | parental satisfaction after 12 months
  1 Very dissatisfied 2 Dissatisfied 3 Neutrally satisfied 4 Satisfied 5 Very satisfied
Child satisfaction Measured immediately post-cementation using a Smiley Face Likert scale in child-friendly language. | immediately after crown cementation
  Child Satisfaction (Smiley Face Likert Scale) awful not very good good really good fantastic

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt

REFERENCES:
- [Background] American Academy of Pediatric Dentistry. Pulp therapy for primary and immature permanent teeth Chicago (IL): American Academy of Pediatric Dentistry; 2023. 2. Abdelwahab DH KN, Badran AS, Darwish D, Abd El Geleel OM. Oneyear radiographic and clinical performance of bioactive materials in primary molar pulpotomy: A randomized controlled trial. J Dent 2024;143:104864. 3. Wang Z. Bioceramic materials in endodontics. Endod Topics 2015;32:3- 30. 4. Mahgoub N, Alqadasi B, Aldhorae K, Assiry A, Altawili ZM, Tao H. Comparison between iRoot BP Plus (EndoSequence Root Repair Material) and Mineral Trioxide Aggregate as Pulp-capping Agents: A Systematic Review. J Int Soc Prev Community Dent 2019;9:542-52. 5. Moazzami F, Sahebi S, Shirzadi S, Azadeh N. Comparative in vitro Assessment of Tooth Color Change under the Influence of Nano Fast Cement and MTA. J Dent (Shiraz) 2021;22:48-52. 6. Ayoub KM, Nagy MM, Aly RM, El Deen GN, El-Batouty K. Effect of Bio MTA plus & ProRoot MTA pulp capping materials on the regenerative properties of human dental pulp stem cells. Sci Rep 2025;15:4749. 7. Voicu G, Didilescu AC, Stoian AB, Dumitriu C, Greabu M, Andrei M. Mineralogical and Microstructural Characteristics of Two Dental Pulp Capping Materials. Materials (Basel) 2019;12:1772. 25 8. Kiranmayi T, Vemagiri CT, Rayala C, Chandrappa V, Bathula H, Challagulla A. In vivo comparison of bioceramic putty and mineral trioxide aggregate as pulpotomy medicament in primary molars. A 12- month follow-up randomized clinical trial. Dent Res J (Isfahan) 2022;19:84. 9. Alqahtani AS, Alsuhaibani NN, Sulimany AM, Bawazir OA. NeoPUTTY(®) Versus NeoMTA 2(®) as a Pulpotomy Medicament for Primary Molars: A Randomized Clinical Trial. Pediatr Dent 2023;45:240-4. 10. Arvelaiz C, Fernandes A, Graterol V, Gomez K, Gomez-Sosa JF, Caviedes-Bucheli J, et al. In Vitro Comparison of MTA and BC RRMFast Set Putty as Retrograde Filling Materials. Eur Endod J 2022;7:203- 9. 11. Motwani N, Ikhar A, Nikhade P, Chandak M, Rathi